CLINICAL TRIAL: NCT04450212
Title: Vitamin K Supplementation Study in Healthy Volunteers (Aim 2B)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds to complete the study.
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Thummel, Professor: Pharmaceutics, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001593; P01GM116691-02S1 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-29 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Vitamin K Status
Keywords: vitamin K; pharmacogenetics; blood clotting factors; CYP4F2
MeSH Terms: interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic; Vitamin K; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: This is a two-phase study. Healthy adults are screened by genetic analysis in phase I and two sub-groups with specific CYP4F2 genotypes (*1/*1 and *1/*3 or *3/*3) are selected to receive vitamin K supplementation in phase II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I, Buccal Swab Collection for DNA Isolation (Experimental): Approximately 200 healthy volunteers recruited. They complete a brief demographic survey and a undergo one-time buccal swab for collection of cheek cells for DNA analysis.
  Interventions: Genetic: Phase I, Buccal Swab Collection for DNA Isolation
- Phase II, Vitamin K (Vitacost) Supplementation (Experimental): Subjects from Phase I with a homozygous CYP4F2*1 (n=14) or CYP4F2*3 carriers (n=14) are selected to receive daily vitamin K supplementation, for 10-days. Blood and urine samples are collected sequentially, at baseline, and during the supplementation period.
  Interventions: Dietary Supplement: Phase II, Vitamin K (Vitacost) Supplementation

INTERVENTIONS:
Genetic: Phase I, Buccal Swab Collection for DNA Isolation — Buccal swab will be taken from study participants for DNA isolation.
  Arms: Phase I, Buccal Swab Collection for DNA Isolation
Dietary Supplement: Phase II, Vitamin K (Vitacost) Supplementation — 1-mg/day phylloquinone (Vitacost; Natures Life K-1 Phylloquinone) for 10 consecutive days. Each dose will be taken in the morning (~ 8 am), with one half pint of 2% milk to facilitate absorption. Blood and urine samples collection before and during the vitamin K supplementation period.
  Arms: Phase II, Vitamin K (Vitacost) Supplementation

SUMMARY:
The overall purpose of this study is to determine how variation in the CYP4F2 gene modulates the synthesis of vitamin K-dependent clotting factors. We propose that the CYP4F2*3 gene variant increases short- and long-term vitamin K concentrations in the liver by reducing the efficiency of vitamin K metabolism. The investigators will study the effect of vitamin K supplementation on two biomarkers of hepatic vitamin K concentration in groups with defined CYP4F2*3 genotype. Specifically, the investigators will test for an association between our novel biomarkers of long-term (plasma Factor II proteoforms) and short-term (urinary K-Acid catabolites) hepatic vitamin K concentration and CYP4F2*3 following a 10-day period of vitamin K supplementation in healthy volunteers.

DETAILED DESCRIPTION:
The investigators will study the effect of vitamin K supplementation on two biomarkers of hepatic vitamin K concentration in groups with defined CYP4F2*3 genotype. Specifically, the investigators will test for an association between our novel biomarkers of long-term (plasma Factor II proteoforms) and short-term (urinary K-Acid catabolites) hepatic vitamin K concentration and CYP4F2*3 following a 10-day period of vitamin K supplementation in healthy volunteers.

The investigators will recruit, by posted advertisements at UWMC, male and female healthy volunteers. A two-step selection process will be employed. Subjects will self-select by responding to flyers, and contact the research coordinator. The research coordinator will screen them for eligibility over the phone and if eligible, make an appointment for the first study visit. For the first phase, the Research Coordinator will collect a buccal swab of DNA from ~ 200 eligible candidates; the DNA will be tested for absence or presence of the CYP4F2*3 variant allele. The PI and Research Coordinator will review the genotyping results and then select 14 individuals with either a homozygous CYP4F2*3 genotype or a heterozygous CYP4F2*1/*3 genotype, and a demographically matched group of 14 with a homozygous CYP4F2*1 genotype at the diagnostic locus for the supplementation phase of the study. The study coordinator will then contact these subjects by phone for Phase II participation.

Procedures - Phase I, Buccal Swab Collection for DNA Isolation.

Demographic Questionnaire: Self-reported heritage, age, and sex will be collected through a brief demographic questionnaire.

Buccal Swab: We will collect cheek cells with a cotton swab and isolate DNA and test for the CYP4F2*1 and CYP4F2*3 alleles.

Genotyping: CYP4F2 genotype will be determined by a validated TaqMan assay (ABI/ThermoFisher Scientific), using commercially available DNA hybridization probes to test for the absence or presence of the CYP4F2*3 allele. Subjects who are either a homozygous CYP4F2*3 genotype or a heterozygous CYP4F2*1/*3 genotype, and CYP4F2*3 alleles will be eligible for Phase II.

Procedures - Phase II, Vitamin K Supplementation.

Vitamin K Supplementation: Research participants selected for the supplementation study based on CYP4F2 genotype will be given 1-mg/day phylloquinone (Vitacost; Natures Life K-1 Phylloquinone) for 10 consecutive days. Each dose will be taken in the morning (~ 8 am), with one half pint of 2% milk to facilitate absorption.

Sample Collection: For the supplementation study, a venous blood sample (10 mL EDTA tube) and a spot urine sample will be collected after an overnight fast from d1 through d5 and on d8 and d10 of Vitamin K supplementation for 10 days. Plasma will be isolated and both samples will be stored at -70°C until analysis. Women of child-bearing potential will have a urine pregnancy test of d1 and if positive, will be withdrawn from the study, and all samples and data will be destroyed.

Measurement of Plasma Factor II Proteoforms: Plasma concentration of the 11 individual proteoforms of Factor II will be measured byLC-MS/MS. This data will be used to calculate three metrics of long-term vitamin K status, unFII, ucFII:iFII and inFII:aFII. These represent different mathematical measures of the degree of Factor II undercarboxylation. Prospective analysis of plasma vitamin K1, PIVKA II and ucOC is not planned, but will be held in reserve should the need for that data arise.

Measurement of Urinary K-Acid I and II: Quantitation of K-Acid I and II, and creatinine (Cr) in spot urine samples will be performed, using a validated LC-MS/MS assay that the investigators have recently developed. The total and individual urinary K-Acid/Cr ratio will be computed.

Statistical Analysis Plan: The investigators will conduct an unpaired t-test to compare the mean response to vitamin K supplementation in the two CYP4F2 genotype groups. Response is defined as the area under the vitamin K status value x time curve, corrected for baseline, for the 10-day intervention period. A secondary metric will be the absolute peak change in the vitamin K status ratio. Both short (urinary K-Acid/Cr ratio) and long-term (ucFII:iFII and inFII:aFII) biomarkers will tested separately. Based on pilot data, a sample size of 14 in each genotype group will provide a power of at least 80% to detect a significant effect at the significance 0.05 level, when there is a two-fold difference in the response to supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be males or females 18 years and older.
2. Participants must read and understand English.
3. Participants must be able to provide informed consent.
4. Women not currently pregnant or lactating.

Exclusion Criteria:

1. Participants less than 18 years of age.
2. Participants unable to read and understand English.
3. Participants unable to provide informed consent.
4. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Short-term Hepatic Vitamin K Status-1 | 10-days
  urinary vitamin K-acid/creatinine ratio
Long-term Hepatic Vitamin K Status | 10-days
  plasma factor II carboxylation state

SECONDARY OUTCOMES:
Short-term Hepatic Vitamin K Status-2 | 10-days
  Plasma vitamin K acid concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Thummel, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No